CLINICAL TRIAL: NCT04978454
Title: A Multicenter, Blinded, Randomized, Placebo-Controlled, Dose-Ranging Influenza Challenge Study in Healthy Adult Volunteers to Determine the Optimal Infection Dose and Safety of a Recombinant H3N2 (A/Texas/71/2017 (H3N2), Clade 3C3a) Influenza Challenge Virus
Brief Title: Influenza Challenge Study to Determine the Optimal Infection Dose and Safety of a Recombinant H3N2 (A/Texas/71/2017 (H3N2, Clade 3C3a) Influenza Strain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: 20-0005; 75N93019C00054
Record Dates: First submitted 2021-07-15; First posted 2021-07-27 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2023-07-25

CONDITIONS: Influenza
Keywords: A/Texas/71/2017; Influenza; Influenza Challenge Study; Recombinant H3N2; Recombinant H3N2 Influenza Strain; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Cohort 1A (Experimental): 10^4 TCID50of recombinant H3N2 (A/Texas/71/2017, clade 3C3a) 1.0 mL (0.5mL per nostril) influenza virus (n=12) and Sham Sucrose phosphate glutamate (SPG) inoculum 1.0 mL (0.5mL per nostril) (n=1) administered intranasally on Day 1. If 80% or more subjects in Cohort 1A meet the case definition for influenza, proceed to Cohort 1B. If fewer than 80% of subjects meet the case definition for influenza in Cohort 1A, the dose will escalate to include Cohort 2A. N = 13
  Interventions: Biological: Influenza RG-A/Texas/71/2017 (H3N2) Challenge; Other: Placebo
- Cohort 1B (Experimental): 10^4 TCID50 of recombinant H3N2 (A/Texas/71/2017, clade 3C3a) 1.0 mL (0.5 mL per nostril) influenza virus (n=12) and Sham Sucrose phosphate glutamate (SPG) inoculum 1.0 mL (0.5 mL per nostril) (n=1) administered intranasally on Day 1. If 80% or more subjects in Cohort 1A and 1B meet the case definition for influenza, proceed to Cohort 1C. Cumulatively, if fewer than 80% of subjects in Cohorts 1A and 1B meet the case definition for influenza, the dose will escalate to include Cohort 2A. N = 13
  Interventions: Biological: Influenza RG-A/Texas/71/2017 (H3N2) Challenge; Other: Placebo
- Cohort 1C (Experimental): 10^4 TCID50 of recombinant H3N2 (A/Texas/71/2017, clade 3C3a) 1.0 mL (0.5 mL per nostril) influenza virus (n=12) and sham sucrose phosphate glutamate (SPG) inoculum 1.0 mL (0.5 mL per nostril) (n=1) administered intranasally on Day 1. If 80% or more of the subjects in Cohorts 1A, 1B, and 1C combined meet the case definition for influenza then the optimal dose of 104 TCID50 will be selected. Cumulatively, if fewer than 80% of subjects in Cohorts 1A, 1B, and 1C meet the case definition for influenza the dose will escalate to include Cohort 2A. N = 13
  Interventions: Biological: Influenza RG-A/Texas/71/2017 (H3N2) Challenge; Other: Placebo
- Cohort 2A (Experimental): 10^5 TCID50 of recombinant H3N2 (A/Texas/71/2017, clade 3C3a) 1.0 mL (0.5 mL per nostril) influenza virus (n=12) and Sham Sucrose phosphate glutamate (SPG) inoculum 1.0 mL (0.5 mL per nostril) (n=1) administered intranasally on Day 1. If 70% or more subjects in Cohort 2A meet the case definition for influenza, proceed to Cohort 1B. If fewer than 70% of subjects meet the case definition for influenza in Cohort 2A, the dose will escalate to include Cohort 3A. N = 13
  Interventions: Biological: Influenza RG-A/Texas/71/2017 (H3N2) Challenge; Other: Placebo
- Cohort 2B (Experimental): 10^5 TCID50 of recombinant H3N2 (A/Texas/71/2017, clade 3C3a) 1.0 mL (0.5 mL per nostril) influenza virus (n=12) and Sham Sucrose phosphate glutamate (SPG) inoculum 1.0 mL (0.5 mL per nostril) (n=1) administered intranasally on Day 1.If 70% or more subjects in Cohort 2A and 2B meet the case definition for influenza, proceed to Cohort 2C. Cumulatively, if fewer than 70% of subjects in Cohorts 2A and 2B meet the case definition for influenza, the dose will escalate to include Cohort 3A N = 13
  Interventions: Biological: Influenza RG-A/Texas/71/2017 (H3N2) Challenge; Other: Placebo
- Cohort 2C (Experimental): 10^5 TCID50 of recombinant H3N2 (A/Texas/71/2017, clade 3C3a) 1.0 mL (0.5 mL per nostril) influenza virus (n=12) and Sham Sucrose phosphate glutamate (SPG) inoculum 1.0 mL (0.5 mL per nostril) (n=1) administered intranasally on Day 1. If 70% or more of the subjects in Cohorts 2A, 2B, and 2C combined meet the case definition for influenza then the optimal dose of 10^4 TCID50 will be selected. Cumulatively, if fewer than 70% of subjects in Cohorts 2A, 2B, and 2C meet the case definition for influenza the dose will escalate to include Cohort 3A. N = 13
  Interventions: Biological: Influenza RG-A/Texas/71/2017 (H3N2) Challenge; Other: Placebo
- Cohort 3A (Experimental): 10^6 TCID50 of recombinant H3N2 (A/Texas/71/2017, clade 3C3a) 1.0 mL (0.5 mL per nostril) influenza virus (n=17) and Sham Sucrose phosphate glutamate (SPG) inoculum 1.0 mL (0.5 mL per nostril) (n=1) administered intranasally on Day 1. If no safety threshold is met (halting conditions) proceed to Cohort 3B. N = 18
  Interventions: Biological: Influenza RG-A/Texas/71/2017 (H3N2) Challenge; Other: Placebo
- Cohort 3B (Experimental): 10^6 TCID50 of recombinant H3N2 (A/Texas/71/2017, clade 3C3a) 1.0 mL (0.5 mL per nostril) influenza virus (n=17) and Sham Sucrose phosphate glutamate (SPG) inoculum 1.0 mL (0.5 mL per nostril) (n=1) administered intranasally on Day 1. N = 18
  Interventions: Biological: Influenza RG-A/Texas/71/2017 (H3N2) Challenge; Other: Placebo

INTERVENTIONS:
Biological: Influenza RG-A/Texas/71/2017 (H3N2) Challenge — RG-A/Texas/71/2017 (H3N2) is an infectious influenza virus and requires handling at BioSafety Level 2. The challenge virus will be administered intranasally in a volume of approximately 0.5 mL per nostril. Intranasal challenge will be carried out using the Intranasal Mucosal Atomization ( MAD Nasa(TM)) Device attached to a 1 mL syringe.
Other: Placebo — Sucrose phosphate glutamate (SPG) inoculum

SUMMARY:
An open-label, dose-ranging influenza challenge study in healthy adult volunteers to determine the optimal infection dose and safety of a recombinant H3N2 (A/Texas/ A/Texas/71/2017 (H3N2, clade 3C3a) influenza strain. The goal of this study is to find a challenge virus dose that is safe and can achieve a symptomatic influenza Attack Rate (AR) that will be sufficiently high for utilization in future vaccine or intervention studies. The optimal dose of the three considered is broadly defined as the minimum challenge virus dose that elicits the highest AR without meeting safety-stopping criteria. Additionally, viral recovery, clinical symptoms, and immune responses over the post-challenge period will be described by challenge dose group. This study will last for up to 1 year depending upon the number of challenge cohorts enrolled given the adaptive dose-escalation design. The populations are healthy males and non-pregnant, non-breastfeeding females aged = 18 and < 46 years of age with a serum HAI antibody titer of </=1:40 against influenza A/Texas/71/2017 (H3N2), clade 3C3a. The study will enroll and challenge up to 106 (plus 8 shams) healthy adult volunteers with the H3N2 (A/Texas/71/2017 (H3N2), clade 3C3a) influenza virus challenge strain. The primary objectives are: 1) To determine the optimal infectious dose of a recombinant influenza virus (A/Texas/71/2017 (H3N2), clade 3C3a) to be used as a clinical challenge strain in future vaccine efficacy or intervention studies as assessed by viral shedding and clinical symptoms. 2) To describe viral detection by quantitative and qualitative Reverse Transcription - Polymerase Chain Reaction (RT-PCR) from study subjects at baseline and post-challenge. 3) To document clinical symptoms from self-reported surveys and standardized symptom scales at baseline and post-challenge.

DETAILED DESCRIPTION:
An open-label, dose-ranging influenza challenge study in healthy adult volunteers to determine the optimal infection dose and safety of a recombinant H3N2 (A/Texas/ A/Texas/71/2017 (H3N2, clade 3C3a) influenza strain. The goal of this study is to find a challenge virus dose that is safe and can achieve a symptomatic influenza Attack Rate (AR) that will be sufficiently high for utilization in future vaccine or intervention studies. The optimal dose of the three considered is broadly defined as the minimum challenge virus dose that elicits the highest AR without meeting safety-stopping criteria. Additionally, viral recovery, clinical symptoms, and immune responses over the post-challenge period will be described by challenge dose group. This study will last for up to 1 year depending upon the number of challenge cohorts enrolled given the adaptive dose-escalation design. The populations are healthy males and non-pregnant, non-breastfeeding females aged = 18 and < 46 years of age with a serum HAI antibody titer of </=1:40 against influenza A/Texas/71/2017 (H3N2), clade 3C3a. The study will enroll and challenge up to 106 (plus 8 shams) healthy adult volunteers with the H3N2 (A/Texas/71/2017 (H3N2), clade 3C3a) influenza virus challenge strain. Subjects will be pre-screened for study inclusion to have serological HAI antibody titers of </=1:40 against the clinical challenge strain. Eligible participants will be enrolled sequentially into dosing cohorts and will be randomly assigned to receive a single dose of either placebo (sham inoculum) or a virus dose between 104 to 106 Median Issue Culture Infectious Dose (TCID50) (in an allocation of 1:12 to 1:17). Dose titration will be conducted under an adaptive escalation schedule whereby dosing will start at the lowest dose 104 TCID50 and only escalate to the next dose if a pre-determined infection and symptomatic attack rate are not met and the dose is determined to be safe and no pre-defined halting rule is met. The attack rate (AR), defined as the percentage of subjects meeting shedding and symptom criteria for symptomatic influenza virus infection (see clinical case definition below), will be determined for each challenge dose group in order to identify the optimal infectious dose (55%-80% AR). This adaptive, dose-ranging approach allows adjustments to challenge dose group size and escalation dose schedule to be informed by the AR and safety results. The primary objectives are: 1) To determine the optimal infectious dose1 of a recombinant influenza virus (A/Texas/71/2017 (H3N2), clade 3C3a) to be used as a clinical challenge strain in future vaccine efficacy or intervention studies as assessed by viral shedding and clinical symptoms. 2) To describe viral detection by quantitative and qualitative Reverse Transcription - Polymerase Chain Reaction (RT-PCR) from study subjects at baseline and post-challenge. 3) To document clinical symptoms from self-reported surveys and standardized symptom scales at baseline and post-challenge. The secondary objectives are: 1) To assess the safety profile of a live recombinant influenza strain (A/Texas/71/2017 (H3N2), clade 3C3a) following challenge in healthy adult volunteers. 2) To describe the host serum hemagglutination inhibition and microneutralization antibody responses at baseline and post-challenge. 3) To describe anti-Hemagglutination(HA)-stalk antibody titer at baseline and post-challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedure
2. Are able to understand and comply with planned study procedures and be available for all study visits
3. Agree to remain an inpatient for at least 7 days after challenge AND until they have no viral shedding*, determined by qualitative Reverse Transcription - Polymerase Chain Reaction (RT-PCR) beginning on Study Day 6

   * No viral shedding is defined as two negative RT-PCR tests 12 or more hours apart
4. Healthy* males and non-pregnant, non-breastfeeding females aged > / = 18 and < 46 years of age at enrollment

   *Healthy is defined in inclusion criteria #11. NOTE: Female subjects of childbearing potential must have a negative serum pregnancy test at screening, a negative urine pregnancy test upon admission to the confinement unit AND a negative pregnancy test before any Chest x-ray (CXR) (if > / = 7 days have passed since a serum pregnancy test).
5. Women of childbearing potential* must agree to use or have practiced true abstinence** or use at least one acceptable primary form of contraception* for at least 30 days prior to challenge

   * Not of childbearing potential - post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, tubal ligation/salpingectomy, or Essure(R) placement with history of documented radiological confirmation test at least 90 days after the procedure).
   * True abstinence is 100% of time no sexual intercourse (male's penis enters the female's vagina). (Periodic abstinence [e.g. calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

     * Acceptable forms of primary contraception include monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the influenza challenge virus, intrauterine devices, birth control pills, and injectable/implantable/insertable hormonal birth control products. Must use at least one acceptable primary form of contraception for at least 30 days prior to challenge and at least one acceptable primary form of contraception during the remainder of the study or approximately 57 days after confinement.

   NOTE: These criteria are applicable to female subjects in a heterosexual relationship AND of child-bearing potential. These criteria do not apply to subjects in a same sex relationship.
6. Non-habitual smoker* of tobacco, e-cigarettes or marijuana

   *Non-habitual smokers are those who smoke no more than four cigarettes, other tobacco products, e-cigarettes (to include vaping and Juuling products) or marijuana in a week and agree not to smoke cigarettes, other tobacco products, e-cigarettes and/or marijuana products during participation in the study.
7. No self-reported or known history of alcoholism within the last 2 years and agrees to abstain from alcohol for at least one week before admission and throughout the confinement period.
8. No self-reported or known history of restricted drug use* for at least 30 days prior to challenge and agrees to abstain from restricted drugs for at least one week before admission and throughout the confinement period
9. Negative drug urine toxicology result on screening (i.e., amphetamines, cocaine, and opiates) and on admission to the confinement unit (i.e., amphetamines, cocaine, and opiates)*

   *Select drug use may be allowed at Investigator's discretion (e.g., prescribed amphetamines for ADHD)
10. Agree not to use the listed prescription or over the counter medications* within 7 days prior to and through confinement period, unless approved by the investigator

    *Oseltamivir, zanamivir, peramivir, baloxavir marboxil, amantadine (generic) and rimantadine (Flumadine and generic), aspirin, intranasal steroids, decongestants, antihistamines, and other non-steroidal anti-inflammatory drugs (NSAIDs)
11. In good health*, and do not have clinically significant medical, psychiatric, chronic or intermittent health conditions including those listed in Exclusion Criteria

    *Good health, as determined by medical history, medication use and physical examination to evaluate ongoing chronic medical or psychiatric diagnoses or conditions, defined as those that have been present for at least 90 days, which would not affect the assessment of the safety of subjects or the immunogenicity of challenge. These medical diagnoses or conditions should be stable for the last 90 days (no hospitalizations, emergency room (ER) or urgent care for condition (excluding musculoskeletal conditions) and not listed in Exclusion Criteria. Subjects may be on medications only if the condition or disease is stable and not deteriorating, if the medical intervention (such as device or medication) was not available during the maximal inpatient period of time, medications are not listed in the Exclusion Criteria and pose no additional risk to subject safety or assessment of adverse events. This also includes no change in prescription medication, dose or frequency as a result of new symptoms or deterioration of the medical diagnosis or condition in the 90 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome (e.g., lowering of the dosage or frequency), as determined by the site principal investigator (PI) or designated clinician licensed to make medical diagnoses and listed on Form FDA 1572, will not be considered a deviation of this inclusion criterion.
12. Vital signs as follows:

    * Pulse is 47 to 99 beats per minute, inclusive
    * Systolic blood pressure is 85 to 139 mmHg, inclusive
    * Diastolic blood pressure is 55 to 89 mmHg, inclusive
    * Saturation of Peripheral Oxygen (SpO2) >/= 95%; Respiratory Rate (RR) </= 18
    * Oral temperature is less than 100.6 degrees Fahrenheit
13. Eligibility laboratory values White Blood Cell (WBC), Absolute Lymphocyte Count, Hemoglobin (Hgb), Platelets (PLTs), Alanine Transaminase (ALT) and Creatinine(Cr) are within acceptable parameters*

    *Labs within normal range or grade 1 abnormalities deemed not clinically significant by a study investigator are considered acceptable
14. Body mass index (BMI) > 18.5 and < 40 kg/m2 at screening
15. Other screening tests Electrocardiogram (ECG) and Chest x-ray(CXR) are within normal reference range or not deemed clinically significant by the Principle Investigator(PI) or appropriate sub-investigator*

    *Designated clinician licensed to make medical diagnoses and listed on the Form FDA 1572
16. Negative test for Human Immunodeficiency Virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV) at screening
17. Negative respiratory virus panel by BIOFIRE(R) FILMARRAY(R) respiratory panel by bioMérieux or by Luminex xTAG(R) on Day -2, and Day -1
18. Negative RT-PCR test for severe acute respiratory syndrome coronavirus 2(SARS-CoV 2) on screening and Day -2
19. Hemagglutination Inhibition Test (HAI) antibody titer </=1:40 against influenza A/Texas/71/2017 (H3N2) at screening
20. Receipt of the recommended number of doses of an (Emergency Use Authorization) EUA authorized or licensed coronavirus disease of 2019 (COVID-19) vaccine product = two weeks prior to confinement

Exclusion Criteria:

1. Presence of self-reported or medically documented significant medical or psychiatric condition(s)*

   *Significant medical or psychiatric conditions include but are not limited to:
   1. Respiratory disease (e.g., chronic obstructive pulmonary disease [COPD], asthma) requiring daily medications [Inhaled, oral or intravenous (IV) corticosteroids, leukotriene modifiers, long and short acting beta agonists, theophylline, ipratropium, biologics] or any treatment for respiratory disease exacerbations (e.g., asthma exacerbation) within the last 5 years
   2. Presence of any febrile illness or symptoms suggestive of a respiratory infection within two weeks prior to challenge
   3. Significant cardiovascular disease (e.g., congestive heart failure, cardiomyopathy, ischemic heart disease) or history of myocarditis or pericarditis as an adult.
   4. Neurological or neurodevelopmental conditions (e.g., epilepsy, stroke, seizures, encephalopathy, focal neurologic deficits, Guillain-Barre syndrome, encephalomyelitis or transverse myelitis).
   5. Ongoing malignancy or recent diagnosis of malignancy in the last five years (excluding basal cell carcinoma of the skin)
   6. Presence of an autoimmune disease.
   7. Immunodeficiency of any cause.
   8. History of diabetes.
2. Presence of immunosuppression or any medications that may be associated with impaired immune responsiveness*

   *Including, but not limited to, corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or systemic corticosteroids or other similar or toxic drugs during the preceding 12-month period prior to screening. Low dose topical and intranasal steroid preparations used for a discrete period of time are permitted.
3. Known allergy or intolerance to treatments for influenza (including any neuraminidase inhibitors or baloxavir marboxil).
4. Known allergy to two or more classes of antibiotics (e.g., penicillins, cephalosporins, fluoroquinolones, or glycopeptides).
5. Known allergy to excipients* in the challenge virus inoculum.

   *Sucrose, KH2PO4, K2HPO4, L-glutamic acid (in SPG diluent)
6. Receipt or planned receipt of any investigational drug/investigational vaccine/licensed vaccine, except for a licensed or emergency use authorized coronavirus disease of 2019 (COVID-19) vaccine product, within 30 days prior to the date of challenge.
7. Prior enrollment in an influenza virus challenge study with an influenza virus of the same subtype within the past 2 years.
8. Currently enrolled in any investigational study or intends to enroll in such a study within the ensuing study period.*

   *Co-enrollment in an observational study, an investigational study in a follow-up/post-vaccination stage, or a study involving a licensed drug or biologic may be allowed at the investigator's discretion.
9. Receipt of any influenza vaccine four months prior to challenge or plans to receive influenza vaccine during the study (approximately 57 days after challenge).
10. History of a previous severe allergic reaction to any drug or biologic with generalized urticaria, angioedema, or anaphylaxis.
11. Receipt of blood or blood products during the six months prior to the planned date of challenge.
12. Plans to donate blood or blood products during the study. (approximately 102 days).
13. Any condition (including medical and psychiatric conditions) that, in the opinion of the Investigator, might interfere with the safety of the subject and/or study objectives.
14. An ongoing symptomatic condition for which subject has had or has ongoing medical investigations but has not yet received a diagnosis or treatment plan e.g., ongoing fatigue without a diagnosis.
15. Known close contact with anyone known to have or suspected to have a respiratory viral illness within 7 days prior to challenge.
16. Significant abnormality altering anatomy of nose/nasopharynx (including significant nasal polyps), clinically significant nasal deviation, or nasal/sinus surgery within 180 days prior to challenge.
17. History in the last five years of chronic or frequent intermittent sinusitis.
18. Recent history (180 days) of epistaxis or anatomic or neurologic abnormality impairing the gag reflex or contributing to aspiration.
19. Currently using an internal cardiac device such as a pacemaker or other implanted electronic medical devices.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland, School of Medicine, Center for Vaccine Development and Global Health, Baltimore, Maryland
  - Duke University Trent Drive, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adult volunteers meeting all protocol-defined eligibility criteria. Participants were recruited from the existing cohort that were pre-screened for influenza antibody titers in the screening protocol DMID 20-0004, as well as from other existing participant registries, through advertising, and by word of mouth. Enrollment occurred between 19AUG2021 and 21JUL2022.
Groups:
- 10^4 TCID50 Challenge Virus: Cohort 1A: Participants were intranasally administered 1.0 mL (0.5mL per nostril) of 10^4 TCID50 of recombinant H3N2 (A/Texas/71/2017 (H3N2), clade 3C3a) influenza virus on Day 1.
  Cohorts 1B and 1C were not enrolled; after review by the Internal Safety Review Committee (ISRC), enrollment continued into Cohort 2A.
- 10^5 TCID50 Challenge Virus: Cohort 2A: Participants were intranasally administered 1.0 mL (0.5mL per nostril) of 10^5 TCID50 of recombinant H3N2 (A/Texas/71/2017 (H3N2), clade 3C3a) influenza virus on Day 1.
  Cohorts 2B and 2C were not enrolled; after review by the Internal Safety Review Committee (ISRC), enrollment continued into Cohort 3A.
- 10^6 TCID50 Challenge Virus: Cohorts 3A and 3B: Participants were intranasally administered 1.0 mL (0.5mL per nostril) of 10^6 TCID50 of recombinant H3N2 (A/Texas/71/2017 (H3N2), clade 3C3a) influenza virus on Day 1.
- Sham Inoculum: From Cohorts 1A, 2A, 3A, and 3B: Participants were intranasally administered 1.0 mL (0.5mL per nostril) of sham sucrose phosphate glutamate (SPG) inoculum on Day 1.
Period: Overall Study
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Started | 12 | 10 | 36 | 2
Completed | 12 | 10 | 36 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum | Total
Number analyzed (Participants) | 12 | 10 | 36 | 2 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (5.8) | 37.8 (6.5) | 31.0 (6.0) | 30.5 (2.1) | 32.7 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 13 | 1 | 26
  Male | 7 | 3 | 23 | 1 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 8 | 0 | 10
  Not Hispanic or Latino | 12 | 8 | 28 | 2 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 14 | 0 | 20
  White | 8 | 6 | 18 | 2 | 34
  More than one race | 1 | 0 | 3 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 10 | 36 | 2 | 60
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.08 (4.41) | 30.07 (5.99) | 28.24 (4.36) | 23.80 (0.85) | 27.97 (4.74)

OUTCOME MEASURES:

1. Primary Outcome: Number and Percentage of Participants With Symptomatic Influenza Virus Infection After Challenge.
Description: Symptomatic influenza virus infection is defined as meeting both of the following criteria:
  1. Viral shedding (as determined by a positive qualitative RT-PCR result or a detectable quantitative RT-PCR result) on at least two days beginning 24 hours after challenge until Study Day 8.
  2. A cumulative symptom score = 6 from daily component symptoms computed across any consecutive 5-day window through Day 8 beginning on Day 2 post challenge using a Modified Jackson Score (MJS). MJS ranges from 0 to 36, with higher scores corresponding to worse outcomes.
Time Frame: Day 2 through Day 8
Population: The Safety population consists of all participants who received study influenza challenge or sham inoculum.
Measure: Count of Participants; unit: Participants
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 36 | 2
Participants | 4 | 5 | 28 | 0

2. Primary Outcome: Number and Percentage of Participants With Detected Viral Shedding in Nasopharyngeal (NP) Swabs Each Day Post-challenge.
Description: Viral shedding status (yes/no) is determined by at least one of: a positive qualitative reverse transcription-polymerase chain reaction (RT-PCR) result from multiplex assay, or a detectable quantitative RT-PCR result.
Time Frame: Day 1 through discharge from the inpatient unit (Day 8 to Day 10)
Population: The Safety population consists of all participants who received study influenza challenge or sham inoculum.
Measure: Count of Participants; unit: Participants
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 36 | 2
Participants
  Day 1 | 0 | 0 | 0 | 0
  Day 2 | 4 | 4 | 34 | 0
  Day 3: number analyzed (Participants) | 12 | 10 | 36 | 1
  Day 3 | 2 | 6 | 32 | 0
  Day 4: number analyzed (Participants) | 12 | 10 | 35 | 2
  Day 4 | 3 | 7 | 29 | 0
  Day 5: number analyzed (Participants) | 12 | 10 | 35 | 2
  Day 5 | 5 | 7 | 23 | 0
  Day 6: number analyzed (Participants) | 12 | 10 | 35 | 2
  Day 6 | 4 | 5 | 15 | 0
  Day 7: number analyzed (Participants) | 12 | 9 | 35 | 2
  Day 7 | 3 | 5 | 12 | 0
  Day 8+: number analyzed (Participants) | 12 | 10 | 35 | 2
  Day 8+ | 3 | 2 | 7 | 0

3. Primary Outcome: Mean Peak Viral Load (VL) After Challenge
Description: The magnitude of viral shedding is measured via quantitative RT-PCR. Peak VL post-challenge is computed for each participant as the maximum log-10 viral copies/mL.
Time Frame: Day 2 through Day 8
Population: The Safety population consists of all participants who received study influenza challenge or sham inoculum. This analysis includes all participants in the Safety population who completed the inpatient period.
Measure: Mean (95% Confidence Interval); unit: log-10 viral copies/mL
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 35 | 2
log-10 viral copies/mL | 1.2154 [0.1236 to 2.4036] | 2.6931 [1.3234 to 4.0380] | 2.6570 [2.1464 to 3.1694] | NA [NA to NA] — All participants in the Sham Inoculum group did not exhibit any quantitative RT-PCR results at or above the lower limit of detection for the assay.

4. Primary Outcome: Mean Duration of Viral Shedding
Description: Viral shedding status (yes/no) for each day during the challenge period is determined by at least one of: a positive qualitative RT-PCR result from multiplex assay, or a detectable quantitative RT-PCR result. The duration of shedding for each participant was computed as the number of days from the initial positive NP swab until the day after the final positive NP swab. Intermittent negative results were ignored for this computation.
Time Frame: Day 2 through Day 8
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 35 | 2
days | 2.3 [0.9 to 4.0] | 3.8 [2.1 to 5.3] | 4.4 [3.8 to 5.1] | NA [NA to NA] — All participants in the Sham Inoculum group did not exhibit any quantitative RT-PCR results at or above the lower limit of detection for the assay.

5. Primary Outcome: Mean Maximum Cumulative Modified Jackson Score (MJS)
Description: The cumulative symptom score from daily component symptoms is computed across any consecutive 5-day window through Day 8 beginning on Day 2 post challenge using the Modified Jackson Score (MJS). MJS ranges from 0 to 36, with higher scores corresponding to worse outcomes. The maximum cumulative score post-challenge was computed for each participant.
Time Frame: Day 2 through Day 8
Population: The Safety population consists of all participants who received study influenza challenge or sham inoculum.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 36 | 2
score on a scale | 13 [6.4 to 21.2] | 15.9 [7.2 to 25.4] | 25.8 [18.3 to 34.1] | 1.0 [NA to NA] — A confidence interval could not be calculated due to all participants having the same maximum score.

6. Primary Outcome: Number and Percentage of Participants Symptomatic for Influenza.
Description: Participants were categorized as symptomatic if they reported a cumulative symptom score = 6 from daily component symptoms computed across any consecutive 5-day window through Day 8 beginning on Day 2 post challenge using a Modified Jackson Score (MJS). MJS ranges from 0 to 36, with higher scores corresponding to worse outcomes.
Time Frame: Day 2 through Day 8
Population: The Safety population consists of all participants who received study influenza challenge or sham inoculum.
Measure: Count of Participants; unit: Participants
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 36 | 2
Participants | 8 | 6 | 29 | 0

7. Secondary Outcome: Number of Adverse Events (AEs) Reported From Challenge Through Day 29
Description: Adverse events were defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product. Non-serious, unsolicited adverse events were collected from Day 1 through Day 29. Serious adverse events were collected from Day 1 through Day 57. Adverse events were MedDRA coded.
Time Frame: Day 1 through Day 29
Population: The Safety population consists of all participants who received study influenza challenge or sham inoculum.
Measure: Number; unit: events
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 36 | 2
events | 10 | 16 | 28 | 3

8. Secondary Outcome: Number and Percentage of Participants Reporting Any AE From Challenge Through Day 29.
Description: as for outcome 7
Time Frame: Day 1 through Day 29
Population: The Safety population consists of all participants who received study influenza challenge or sham inoculum.
Measure: Count of Participants; unit: Participants
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 36 | 2
Participants | 6 | 8 | 17 | 2

9. Secondary Outcome: Number of Serious Adverse Events (SAEs) Reported From Challenge Through Day 57
Description: An adverse event or suspected adverse reaction is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Day 1 through Day 57
Population: The Safety population consists of all participants who received study influenza challenge or sham inoculum.
Measure: Number; unit: events
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 36 | 2
events | 0 | 0 | 0 | 0

10. Secondary Outcome: Number and Percentage of Participants Reporting an SAE at Any Time From Challenge Through Day 57
Description: as for outcome 9
Time Frame: Day 1 through Day 57
Population: The Safety population consists of all participants who received study influenza challenge or sham inoculum.
Measure: Count of Participants; unit: Participants
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 36 | 2
Participants | 0 | 0 | 0 | 0

11. Secondary Outcome: Number and Percentage of Participants With Serological Conversion for Hemagglutination Inhibition (HAI) Antibody Titers Against A/Texas/71/2017 (H3N2), Clade 3C3a Virus, by Study Day
Description: Serological conversion (seroconversion) is defined as a minimum 4-fold rise in post-challenge antibody titers, compared to baseline. Titers for each participant are estimated as the geometric mean of technical replicate results, and the geometric mean is taken again across participants in each challenge dose group.
Time Frame: Day 8, Day 15, and Day 29
Population: The Intent-to-Treat population consists of all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 35 | 2
Participants
  Day 8 | 0 | 1 | 4 | 0
  Day 15 | 2 | 4 | 14 | 0
  Day 29: number analyzed (Participants) | 11 | 10 | 35 | 2
  Day 29 | 1 | 4 | 14 | 0

12. Secondary Outcome: Geometric Mean Hemagglutination Inhibition (HAI) Antibody Titers Against A/Texas/71/2017 (H3N2), Clade 3C3a Virus, by Study Day
Description: Titers for each participant are estimated as the geometric mean of technical replicate results, and the geometric mean is taken again across participants in each challenge dose group.
Time Frame: Day -1 (baseline), Day 8, Day 15, and Day 29
Population: The Intent-to-Treat population consists of all enrolled participants.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 36 | 2
titer
  Day -1 | 10.9 [7.3 to 16.8] | 7.6 [5.4 to 10.7] | 10.7 [8.4 to 13.9] | 5.0 [NA to NA] — A confidence interval could not be calculated due to all participants having the same geometric mean titer.
  Day 8 | 11.2 [7.9 to 16.3] | 8.7 [5.7 to 14.1] | 15.9 [11.6 to 21.9] | 5.0 [NA to NA] — A confidence interval could not be calculated due to all participants having the same geometric mean titer.
  Day 15 | 25.2 [17.8 to 37.8] | 36.1 [21.4 to 65.0] | 37.0 [28.9 to 47.3] | 5.0 [NA to NA] — A confidence interval could not be calculated due to all participants having the same geometric mean titer.
  Day 29 | 25.7 [18.8 to 37.6] | 32.5 [17.4 to 65.0] | 33.8 [26.4 to 43.3] | 5.0 [NA to NA] — A confidence interval could not be calculated due to all participants having the same geometric mean titer.

13. Secondary Outcome: Number and Percentage of Participants With Serological Conversion for Microneutralization (MN) Antibody Titers Against A/Texas/71/2017 (H3N2), Clade 3C3a Virus, by Study Day
Description: as for outcome 11
Time Frame: Day 8, Day 15, and Day 29
Population: The Intent-to-Treat population consists of all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 35 | 2
Participants
  Day 8 | 0 | 0 | 5 | 0
  Day 15 | 4 | 7 | 17 | 0
  Day 29: number analyzed (Participants) | 11 | 10 | 35 | 2
  Day 29 | 3 | 6 | 17 | 0

14. Secondary Outcome: Geometric Mean Microneutralization (MN) Antibody Titers Against A/Texas/71/2017 (H3N2), Clade 3C3a Virus, by Study Day
Description: as for outcome 12
Time Frame: Day -1 (baseline), Day 8, Day 15, and Day 29
Population: The Intent-to-Treat population consists of all enrolled participants
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 36 | 2
titer
  Day -1 | 29.1 [17.8 to 46.2] | 16.2 [9.0 to 30.3] | 24.0 [17.8 to 32.4] | 14.1 [10.0 to 20.0]
  Day 8: number analyzed (Participants) | 12 | 10 | 35 | 2
  Day 8 | 37.8 [25.9 to 55.0] | 28.3 [18.7 to 42.9] | 46.9 [35.9 to 61.2] | 23.8 [20.0 to 28.3]
  Day 15: number analyzed (Participants) | 12 | 10 | 35 | 2
  Day 15 | 69.2 [51.9 to 89.8] | 102.0 [77.3 to 139.3] | 85.7 [69.6 to 106.6] | 20.0 [10.0 to 40.0]
  Day 29: number analyzed (Participants) | 11 | 10 | 35 | 2
  Day 29 | 64.2 [46.8 to 85.2] | 82.8 [60.6 to 121.3] | 75.4 [61.8 to 91.9] | 14.1 [10.0 to 20.0]

15. Secondary Outcome: Number and Percentage of Participants With Serological Conversion for HA-stalk-specific Antibody Titers Against A/Texas/71/2017 (H3N2), Clade 3C3a Virus, by Study Day
Description: Serological conversion (seroconversion) is defined as a minimum 4-fold rise in post-challenge antibody titers against HA group 2 stem domains, compared to baseline. Titers for each participant are estimated as the geometric mean of technical replicate results, and the geometric mean is taken again across participants in each challenge dose group.
Time Frame: Day 8, Day 15, and Day 29
Population: The Intent-to-Treat population consists of all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 35 | 2
Participants
  Day 8 | 0 | 2 | 0 | 0
  Day 15 | 1 | 3 | 2 | 0
  Day 29: number analyzed (Participants) | 11 | 10 | 35 | 2
  Day 29 | 0 | 2 | 2 | 0

16. Secondary Outcome: Geometric Mean HA-stalk-specific Antibody Titers Against A/Texas/71/2017 (H3N2), Clade 3C3a Virus, by Study Day
Description: as for outcome 12
Time Frame: Day -1 (baseline), Day 8, Day 15, and Day 29
Population: The Intent-to-Treat population consists of all enrolled participants
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
Number analyzed (Participants) | 12 | 10 | 36 | 2
titer
  Day -1 | 9407.9 [6396.7 to 13735.7] | 5722.8 [3208.0 to 9760.5] | 7938.6 [6028.5 to 10400.8] | 7954.3 [3656.0 to 17306.0]
  Day 8: number analyzed (Participants) | 12 | 10 | 35 | 2
  Day 8 | 9175.2 [6745.1 to 12854.5] | 8904.9 [6836.9 to 11598.0] | 10506.4 [8030.6 to 13663.3] | 7752.2 [3773.0 to 15928.0]
  Day 15: number analyzed (Participants) | 12 | 10 | 35 | 2
  Day 15 | 11227.9 [8286.4 to 15986.4] | 19814.9 [11567.4 to 34824.7] | 14693.3 [11188.6 to 19221.9] | 9238.5 [4573.0 to 18664.0]
  Day 29: number analyzed (Participants) | 11 | 10 | 35 | 2
  Day 29 | 10964.6 [8047.9 to 15552.9] | 16736.1 [9697.6 to 29895.4] | 13989.0 [10715.9 to 18491.2] | 7927.4 [3906.0 to 16089.0]

ADVERSE EVENTS:
Time Frame: Non-serious, unsolicited adverse events were collected from Day 1 through Day 29. Serious adverse events and all-cause mortality were collected from Day 1 through Day 57.
Arm/Group | 10^4 TCID50 Challenge Virus | 10^5 TCID50 Challenge Virus | 10^6 TCID50 Challenge Virus | Sham Inoculum
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10 | 0/36 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10 | 0/36 | 0/2
Other Adverse Events (participants affected / at risk) | 6/12 | 8/10 | 17/36 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10^4 TCID50 Challenge Virus (N=12) | 10^5 TCID50 Challenge Virus (N=10) | 10^6 TCID50 Challenge Virus (N=36) | Sham Inoculum (N=2)
Tachycardia (Cardiac disorders) | 0 (0) | 4 (4) | 3 (3) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (2) | 4 (5) | 0 (0)
Heart rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory rate decreased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Respiratory rate increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/54/NCT04978454/Prot_001.pdf
  • Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/54/NCT04978454/SAP_002.pdf
  • Informed Consent Form (2022-07-08): https://cdn.clinicaltrials.gov/large-docs/54/NCT04978454/ICF_000.pdf